CLINICAL TRIAL: NCT01745354
Title: Intratumoral Injection of an Immunostimulatory CpG, SD-101, Combined With Local Radiation for the Treatment of Recurrent or Progressive Lymphoma After Allogeneic Hematopoietic Cell Transplantation
Brief Title: Immunostimulatory CpG SD-101 + RT in Recurrent/Progressive Lymphoma After Allogeneic Hematopoietic Cell Transplantation (HCT)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Accrual issues - Slow accrual
Sponsor: Robert Lowsky (Other)
Responsible Party: Sponsor-Investigator, Robert Lowsky, Associate Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT235; SU-07212011-8129 (Other: Stanford University); 20741 (Other: stanford IRB)
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Lymphoma, Non-Hodgkin; Hodgkin Disease
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SD-101 + Combined with Local Radiation (Experimental)
  Interventions: Drug: SD-101; Radiation: Local Radiation

INTERVENTIONS:
Drug: SD-101 — SD-101 will be administered after radiation to only the largest palpable lymph node as an intratumoral injection weekly for 3 weeks at three dosing cohorts: 0.3 mg, 1 mg, and 3 mg
  Other Names: Dynavax
Radiation: Local Radiation

SUMMARY:
For patients with lymphoma that recurs after chemotherapy, bone marrow transplantation using cells from a healthy donor represents potentially curative treatment. In these individuals, cure is possible because transplantation of healthy donor immune cells can fight the lymphoma in the patient. The goal of this work is to test a strategy that activates the healthy donor immune cells so that they more effectively fight lymphoma and can result in an increased cure rate for these patients. Our group has previously studied CpG, an immune activating medication, in patients with lymphoma and demonstrated modest anti-tumor responses. We now have a more potent form of CpG which we intend to test to see if it will better activate the donor immune cells and result in shrinkage of tumor throughout the entire body, not just at the injected site.

DETAILED DESCRIPTION:
Patients will receive low dose radiation to all bulky or symptomatic lymph nodes on days -2 and -1. SD-101 will be administered intratumorally to the single largest palpable node within 24 hours after completion of radiation, on day 0. Two additional intratumoral SD-101 injections will be performed on days 7 (+/- 2 days) and 14 (+/- 2 days). This is a dose ranging study using a 3+3 design with a definition of maximum tolerated dose (MTD) which our group has found acceptable in the past. The first cohort of patients will receive a SD-101 dose of 0.3 mg per injection. The dose will be escalated to 1 mg and 3 mg based on dose limiting toxicity (DLT).

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-confirmed relapsed, refractory, or progressive NHL or HL (Refer to Section 3.2.1 for excluded subtypes)
* At least 3 sites of disease

  1. One for diagnosis (lymph node or bone marrow biopsy)
  2. One palpable for treatment
  3. One measurable radiographically
* > 60 days after RIC allogeneic transplant for lymphoma
* 18 years of age or older
* Mixed (5-95%) or complete (>95%) chimerism
* Eastern Oncology Cooperative Group (ECOG) performance status ≤ 2
* ANC >1000/mm3, platelets >50,000/mm3
* Total bilirubin ≤ 2.5 mg/dL, AST and ALT < 3 times upper limit of normal
* Serum creatinine ≤ 3 mg/dL
* No chemotherapy, RT, DLI or biologic therapy for lymphoma at least 4 weeks prior to scheduled treatment
* Minimal immunosuppression (defined as monotherapy with ≤ 10 mg prednisone daily, ≤ 200 mg cyclosporine daily, or ≤ 2 mg tacrolimus daily) at least 2 weeks prior to scheduled treatment

Exclusion Criteria:

* HIV associated lymphoma
* Acute GVHD at time of enrollment (history of treated and resolved GVHD is permitted)
* Active infection within 14 days prior to scheduled treatment
* Active Cytomegalovirus (CMV) disease at the time of enrollment
* Pre-existing autoimmune or antibody mediated disease (including systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, and autoimmune thrombocytopenia)
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Determination of the maximum tolerated dose based on dose limiting toxicity defined as any new grade 3-4 toxicity after the first SD-101 administration | 60 Days

SECONDARY OUTCOMES:
Measure cytotoxic T-cell activity changes pre- and post-treatment of tumor infiltrating lymphocytes and peripheral blood lymphocytes using ELISA and Immunohistochemistry. | 2, 3, 8 weeks after treatment
Measure tumor response by PET-CT scan imaging | 8 weeks after treatment
Measure level of donor specific tumor infiltrating lymphocytes by flow cytometry and Immunofluorescence | 2, 3, 8 weeks after treatment
  Collect PBMCs

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lowsky, Principal Investigator — Stanford University; Lauren Maeda, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States